CLINICAL TRIAL: NCT05899842
Title: Routine Versus Symptomatic Protein Pump Inhibitor Therapy for Prevention of Gastroesophageal Reflux After Per Oral Endoscopic Myotomy for Esophageal Achalasia. Randomized Open-label Clinical Trial
Brief Title: Routine Versus Symptomatic Protein Pump Inhibitor Therapy for Prevention of Gastroesophageal Reflux After Per Oral Endoscopic Myotomy for Esophageal Achalasia
Acronym: IPPOEM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AOIGCSMERRI/2020/LC-01
Record Dates: First submitted 2023-06-02; First posted 2023-06-12 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Esophageal Achalasia
MeSH Terms: conditions — Esophageal Achalasia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Systematic protein pump inhibitor therapy (Experimental)
  Interventions: Drug: Protein pump inhibitor therapy systematically
- Protein pump inhibitor therapy as necessary (No Intervention)

INTERVENTIONS:
Drug: Protein pump inhibitor therapy systematically — Lansoprazole 30mg once per day
  Arms: Systematic protein pump inhibitor therapy

SUMMARY:
Per Oral Endoscopic Myotomy (POEM) is a treatment of choice for achalasia with an excellent safety and efficacy profile. There is a high rate of esophagitis related to gastroesophageal reflux following this procedure. There is no recommendation on the prescription of protein pump inhibitors (PPI) after the procedure and no study has studied the benefit of systematic prescription of PPI after POEM for achalasia. The study authors hypothesize that routine PPI prescribing post-POEM for 12 months would reduce the rate of esophageal acid exposure compared to a symptom-based prescribing strategy.

ELIGIBILITY:
Inclusion Criteria:

* Patient with an indication for esophageal POEM for achalasia
* Patient with all types of achalasia with Eckardt score > 3
* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan

Exclusion Criteria:

* Patient with contraindications to PPIs
* Patient with mediastinal and esophageal neoplasia
* Patient with a history of Heller myotomy surgery
* Patients requiring any type of anti-reflux valve surgery
* The subject is in a period of exclusion determined by a previous study
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* Patient is pregnant, parturient or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Presence of pathological acid reflux between groups | Month 6
  According to the Lyon 2018 criteria: Esophagitis grade C or D according to the Los Angeles classification and/or acid exposure >6% on 24-hour esophageal pH-metry

SECONDARY OUTCOMES:
Presence of pathological acid reflux between groups | Month 12
  According to the Lyon 2018 criteria: Esophagitis grade C or D according to the Los Angeles classification and/or acid exposure >6% on 24-hour esophageal pH-metry
Patient quality of life between groups | Week 6
  WHOQOL-BREF questionnaire
Patient quality of life between groups | Month 6
  WHOQOL-BREF questionnaire
Patient quality of life between groups | Month 12
  WHOQOL-BREF questionnaire
Patient health-related quality of life between groups | Week 6
  Gastroesophageal Reflux Disease Health Related Quality of Life scale (GERD-HRQL)
Patient health-related quality of life between groups | Month 6
  Gastroesophageal Reflux Disease Health Related Quality of Life scale (GERD-HRQL)
Patient health-related quality of life between groups | Month 12
  Gastroesophageal Reflux Disease Health Related Quality of Life scale (GERD-HRQL)
Quantity of PPI consumed between groups | Month 3
  Number of boxes of Lansoprazole consumed as recorded in PPI logbook
Quantity of PPI consumed between groups | Month 6
  Number of boxes of Lansoprazole consumed as recorded in PPI logbook
Quantity of PPI consumed between groups | Month 12
  Number of boxes of Lansoprazole consumed as recorded in PPI logbook
Treatment tolerance between groups | Month 12
  Occurrence of adverse events as recorded by the doctor during patient interview using a scale of Grade 1 (minor) to Grade 5 (death)
Achalasia symptoms between groups | Week 6
  Measured as Eckardt score >3 (score ranging from 0 (no symptoms)-12 (maximum symptoms))
Achalasia symptoms between groups | Month 6
  Measured as Eckardt score >3 (score ranging from 0 (no symptoms)-12 (maximum symptoms))
Achalasia symptoms between groups | Month 12
  Measured as Eckardt score >3 (score ranging from 0 (no symptoms)-12 (maximum symptoms))
Pyrosis symptoms between groups | Month 6
  Classified according to Rome IV criteria: Acid Reflux, Esophageal Hypersensitivity, Functional Pyrosis, Normal
Pyrosis symptoms between groups | Month 12
  Classified according to Rome IV criteria: Acid Reflux, Esophageal Hypersensitivity, Functional Pyrosis, Normal
Patient quality of life between groups | Inclusion
  WHOQOL-BREF questionnaire
Patient health-related quality of life between groups | Inclusion
  Gastroesophageal Reflux Disease Health Related Quality of Life scale (GERD-HRQL)

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Debourdeau, Principal Investigator — CHU de Nimes
Locations (4):
- France (4):
  - AP-HM, Marseille
  - CHU de Montpellier, Montpellier
  - Clinique mutualiste Beausoleil, Montpellier
  - CHU de Nîmes, Nîmes